CLINICAL TRIAL: NCT03798392
Title: A Randomized Comparison of Self-pressurized Air-Q With Blocker With Baska Mask Supraglottic Airway in Low Risk Female Patients Undergoing Ambulatory Surgery.
Brief Title: Self-pressurised Air-Q With Blocker Versus Baska Mask in Low Risk Female Patients Undergoing Ambulatory Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU and pain management - kasr Aiainy Faculty of Medicine - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N-24- 2018
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Supraglottic Airway Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SP group (Active Comparator)
  Interventions: Device: Self-pressurizing Air Q blocker mask measuring airway seal pressure of studied supra-glottic airway devices 10 minutes after insertion
- Baska group (Active Comparator)
  Interventions: Device: Baska mask measuring airway seal pressure of studied supra-glottic airway devices 10 minutes after insertion

INTERVENTIONS:
Device: Self-pressurizing Air Q blocker mask measuring airway seal pressure of studied supra-glottic airway devices 10 minutes after insertion — comparing the airway seal pressure 10 min after insertion of each devices .
  Other Names: airway management under general anesthesia
  Arms: SP group
Device: Baska mask measuring airway seal pressure of studied supra-glottic airway devices 10 minutes after insertion — comparing the airway seal pressure 10 min after insertion of each devices .
  Other Names: airway management under general anesthesia
  Arms: Baska group

SUMMARY:
Supraglottic airway devices (SGAs) are very commonly used during anesthesia but structural vulnerability to airway morbidity and issues about cuff pressure still concern anesthesiologists. There have been controversial results regarding optimal intra-cuff pressure in various types of cuffed supraglottic airways. When the supraglottic cuff pressure is more than the mucosal perfusion pressure, it is likely to either cause postoperative pharyngo-laryngeal symptoms like sore throat (dysphagia, dysphonia) or cause local mucosal trauma and nerve injuries. Supraglottic airway devices with non-inﬂatable cuff have advantages in omitting the cuff pressure monitoring and reducing potential pharyngo-laryngeal complications.

Self-pressurizing Air Q blocker is the latest version. It has a drain tube through which a suction tube is passed. There is an inflatable cuff at the end of this tube. On inflation, the cuff seals the esophageal opening into the stomach, preventing any regurgitation of stomach contents. Instead of the pilot balloon and inﬂating cuff, the air-Q SP with blocker has a communication oriﬁce at the junction of the peri-glotic cuff and the airway tube. This communication between two spaces enables the cuff to dynamically regulate intra-cuff pressure depending on airway pressure. This distinguishing feature of the air-Q SP may result in reduced risk for airway morbidities related to cuff hyperinﬂation.

The Baska mask is a novel supraglottic airway device with a non-inﬂatable cuff, an oesophageal drainage inlet and side channels to facilitate aspiration of gastric contents, and an integrated bite-block. It was revealed that the baska mask is relatively easy to insert, provided a high-quality seal with the glotic aperture and the incidence of throat discomfort appeared low.

To our knowledge, and after searching in previous literature, no previous studies have compared the Air-Q SP with blocker with Baska mask; another supraglottic airway devices with non-inﬂatable cuff.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the age group of 18 and 50 years,
* ASA class I and II,
* undergoing elective surgeries,
* with Ganzouri airway score less than 4

Exclusion Criteria:

* ASA III - V patients.
* Airway score ≥ 4 according to El-Ganzouri Airway Scoring System.
* Patients with respiratory or pharyngeal pathology.
* Patients allergic to any drugs in the protocol.
* Obese patients with body mass index ≥ 40.
* Patients known to have risk of gastric aspiration, gastro-esophageal reflux disease, hiatus hernia or previous upper gastrointestinal tract surgery.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
airway seal pressure 10 minutes after insertion | 10 minutes after the device insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Faculty of Medicine - Cairo university, Cairo, Egypt